CLINICAL TRIAL: NCT00385749
Title: Right Ventricular Defibrillation Lead Select Site Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Associates in Cardiology, PA (Other)
Collaborators: Medtronic (Industry)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RVLeadSelectSite
Record Dates: First submitted 2006-10-10; First posted 2006-10-11 (Estimated); Last update posted 2007-11-01 (Estimated); Status verified 2007-10

CONDITIONS: Heart Failure, Congestive; Tachycardia, Ventricular
Keywords: Implanted cardioverter defibrillator; congestive heart failure; right ventricular lead placement; select site pacing
MeSH Terms: conditions — Heart Failure; Tachycardia, Ventricular

INTERVENTIONS:
Device: RV apical vs RV septal defibrillation threshold testing

SUMMARY:
This study will compare single coil right ventricular defibrillation leads for implanted cardioverter/defibrillators (ICDs) in the apical and high septal locations. It is hypothesized that RV septal positions are at least as good as apical positions using formally measured defibrillation thresholds(DFTs), and that they may have long term advantages in reducing left ventricular dysfunction.

DETAILED DESCRIPTION:
The new studies "Right Ventricular Lead/Select Site Registry" and "Right Ventricular Lead/Select Site Registry: Acute Study" are studies designed to look at alternate lead locations for defibrillation leads for ICDs. The registry is designed to capture data from patients who have already undergone implant, so as to be able to publish long term data on defibrillation thresholds, pacing thresholds and left ventricular function. This will include both patients from the acute study, and those patients in whom leads have already been placed, and the exact lead location is known. The acute study is designed to directly compare defibrillation thresholds in the apical location versus the interventricular septal location for defibrillation leads. This study involves a direct comparison of two different sites in the same patient; using defined criteria for implant location (see protocol). The acute study is anticipated to enroll 34 patients, but the registry to collect ongoing data will be larger, encompassing previously implanted patients, with an expected sample size of 61 total in the registry for data collection.

ELIGIBILITY:
Inclusion Criteria:

* Standard indications for ICD placement (AHA/ACC guidelines)

Exclusion Criteria:

* Inability to consent
* age less than 21 years
* inability to participate in study follow-up

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2006-10; Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
Acute defibrillation thresholds

SECONDARY OUTCOMES:
LV function (LVEF)
pacing thresholds
sensing thresholds
LV diameter
NYHA class
weight

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Lincoln, MD, Principal Investigator — Holy Cross Hospital of Silver Spring
Locations (1):
- Holy Cross Hospital of Silver Spring, Silver Spring, Maryland, United States